CLINICAL TRIAL: NCT04106804
Title: Abatacept Bone Effects in Psoriatic Arthritis With Bone Biomarkers - ABEPSA _ BB
Brief Title: Abatacept Bone Effects in Psoriatic Arthritis With Bone Biomarker
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ABEPSA_BB
Record Dates: First submitted 2019-09-25; First posted 2019-09-27 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Evaluate Bone Changes in Patients With PsA
Keywords: Psoriatic arthritis; Bone
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — Abatacept

STUDY DESIGN:
Intervention Model Description: The study is a single arm interventional study with a treatment phase of 6 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Abatacept 125 MG/ML — Patients will receive weekly abatacept (Orencia®) s.c. Abatacept in the dose regimen given in the label for RA and PsA for six months

SUMMARY:
Observation has pointed out, that osteitis present in the MRI scans, predicts bone erosion and that this in accordance with the concept by underlining the importance of bone marrow involvement in arthritis [Krabben A, 2013]. Abatacept with its favourable safety profile preferentially interrupts activation of naïve T cells and perhaps makes the strongest case for exploiting co-stimulatory blockade during the earliest detectable phase of the adaptive immune response at a time when predisposition to autoimmune disease can be detected.

DETAILED DESCRIPTION:
Psoriatic arthritis (PsA) is a chronic inflammatory arthritis that occurs in individuals with psoriasis. It is estimated that 1% to 3% of the general population have psoriasis.1,2,3 In Europe the prevalence of psoriasis ranges up to 6.5%.4 Between 10% and 30% of subjects with Psoriasis develop arthritis. As a result, PsA is the second most common inflammatory arthropathy, following rheumatoid arthritis (RA). 1,2,3 Psoriatic arthritis, a seronegative spondyloarthropathy, is a complex disease involving peripheral and axial joints and periarticular structures resulting in enthesitis and dactylitis. Without appropriate management, the number of joints affected by PsA and the severity of joint damage increase over time, which can lead to marked restriction of daily activities and to substantially compromised quality of life. There is evidence that active PsA is associated with accelerated atherosclerosis, obesity, metabolic syndrome and cardiovascular disease. Other co-morbidities such as pulmonary fibrosis, uveitis, and, less commonly, aortic insufficiency, also contribute to the complexity of PsA.5 Unlike RA, effective treatment options are limited for PsA. Responses to the traditional disease-modifying anti-rheumatic drugs (DMARDs) have been suboptimal.6 There is a significant unmet medical need for more effective and safe therapies in PsA, especially for reducing the arthritic signs and symptoms as well as inhibiting progression of structural damage in joints. About 20% of subjects with PsA will develop a severe destructive disabling form of arthritis.7 In the absence of definitive therapy, more than 50% of subjects with PsA will develop 5 or more deformed joints within 10 years of the onset of disease.8 TNFi therapies are efficacious for both skin and joint diseases and have been shown to inhibit structural damage, but approximately 40% of subjects treated with TNFi agents do not reach a minimal improvement [American College of Rheumatology [ACR) 20]9,10,11,12.13,14,15,16,17 In addition, serious adverse events (SAEs) including infections and injection site reactions have been associated with the use of TNFi therapies. Although in some studies a small percentage of patients previously exposed to TNFi were included, these studies were not powered to demonstrate efficacy in that sub-population. Thus, in subjects who experience inefficacy or intolerance of TNF blockade, there is still medical need for new options. Therefore, there is still need in PsA for therapies that provide significant improvement in arthritis and a risk benefit profile that is acceptable. Therapies directed at novel targets (IL-12/23, PDE4-Antagonist) are also approved since 2014. 18, 19, 20, 21 Joint involvement, is clearly the most prominent example for the systemic nature of psoriasis. Notably, the burden of joint disease in patients with psoriasis may be even higher, given that not all psoriasis patients experiencing musculoskeletal complaints fulfill the classification criteria of PsA22. If present, PsA is a severe disease associated with impaired function and reduced life quality life.

ELIGIBILITY:
Inclusion Criteria:

* Males/females with CASPAR criteria-positive PsA
* Active disease with more than three swollen and tender joints
* Must be aged ≥ 18 years at time of consent
* ≥ 3 erosions on MRI or HR PQCT
* Women of childbearing potential or men capable of fathering children must be using effective contraception during treatment with abatacept and up to 14 weeks after the last dose of abatacept treatment.
* Must understand and voluntarily sign an informed consent form including written consent for data protection ´- Must be able to adhere to the study visit schedule and other protocol requirements

Exclusion Criteria:

* Previous exposure to abatacept
* CCP2 positivity
* Investigational study drug within 4 weeks (or 5 halflives (half live is 14,3 days), whichever is longer) prior to randomisation
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
* Any other autoimmune or inflammatory disease such as SLE, PSS, MCTD, SpA, Behcet disease, vasculitis or autoimmune hepatitis.
* Any malignancy in the last 5 years
* Chronic infection such as latent TB (TB not adequately treated according to guidelines) or hepatitis B or C infection
* Immunocompromised or HIV-positive patients
* Uncontrolled severe concomitant disease
* Patients who are younger than 18 years or are incapable to understand the aim, importance and consequences of the study and to give legal informed consent (according to § 40 Abs. 4 and § 41 Abs. 2 and Abs. 3 AMG).
* Pregnant or lactating females
* Patients who possibly are dependent on the Principal Investigator or

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-06-06 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Bone Erosion volume | 6 months
  Change in bone erosion volume measured by Hr-PQ CT of the involved hand between baseline and 24 weeks follow-up

SECONDARY OUTCOMES:
Comparing bone Erosion baseline to week 24 | 6 months
  Change in bone erosion on CT between baseline and 24 wks
Comparing Osteophytes between baseline and week 24 | 3 and 6 months
  Change in osteophytes CT between baseline and 24 wks
Comparing Tenosynovitis between baseline, month 3 and month 6 | 3 and 6 months
  Change in MRI Tenosynovitis score between baseline compared to month 3 and 6
Comparing PSAMRIS score between baseline and month 3 and month 6 | 3 and 6 months
  Change in PSAMRIS MRI score between baseline compared to month 3 and 6
Comparing bone Erosion between baseline month 3 and and month 6 with MRI | 3 and 6 months
  Change in MRI bone erosions between baseline compared to month 3 and month 6
Comparing Synovitis between baseline and month 3 and month 6 | 3 and 6 months
  Change in MRI synovitis between baseline compared to month 3 and month 6
Comparing DAS28 from baseline to month 3 and month 6 | 3 and 6 months
  Change of DAS28 between baseline compared to month 3 and month 6
Comparing DAPSA between baseline, month 3 and month 6 | 3 and 6 months
  Change of DAPSA between baseline compared to month 3 and month 6
Comparing MDA from baseline, month 3 and month 6 | 3 and 6 months
  Change of MDA between baseline compared to month 3 and month 6
Comparing HAQ-DI between baseline compared to month 3 and month 6 | 3 and 6 months
  Change of HAQ-DI between baseline compared to month 3 and month 6
Comparing SPARCC between baseline compared to month 3 and month 6 | 3 and 6 months
  Change of SPARCC between baseline compared to month 3 and month 6
Comparing PSAID between baseline compared to month 3 and month 6 | 3 and 6 months
  Change of PSAID between baseline compared to month 3 and month 6
Comparing PASI between baseline compared to month 3 and month 6 | 3 and 6 months
  Change of PASI between baseline compared to month 3 and month 6
Comparing SF36 between screening, month 3 and month 6 | 3 and 6 months
  Change of SF36 between screening, month 3 and month 6

CONTACTS AND LOCATIONS:
Locations (1):
- University Clinic Erlangen, Medical Department 3, Rheumatology & Immunology, Erlangen, Germany

IPD SHARING:
Plan to Share IPD: No